CLINICAL TRIAL: NCT05848063
Title: Effects of Global Hip Versus Isolated Abductors Muscles Strengthening Exerciseprogram on Pain, Range of Motion, and Lower Extremity Function in Patients Withsecondary Piriformis Syndrome
Brief Title: Effects of Global Hip Versus Isolated Abductors Strengthening Exercises in Patients Withsecondary Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0102
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Global hip muscles strengthening exercises (Experimental): Group A Group A will receive hot packs along with all hip muscle strengthening exercises. All exercises were performed for 3 sessions per week for 6 weeks. Outcome measures will be taken at baseline, in 3rd week, and at the end of the 6th week.
  Interventions: Other: Global hip muscles strengthening exercises
- Group B: Hip abductors strengthening exercises (Active Comparator): Group B will receive hot packs along with Hip abductors strengthening. A baseline assessment will be done on eligible participants. 3 sessions were given 3 days per week, Outcome measures will be taken at baseline, in 3rd week, and at the end of the 6th week.
  Interventions: Other: Hip abductors strengthening exercises

INTERVENTIONS:
Other: Global hip muscles strengthening exercises — Strengthening exercises will be given to all hip muscles
  Arms: Group A: Global hip muscles strengthening exercises
Other: Hip abductors strengthening exercises — Strengthening exercises will be given to hip abductor muscles
  Arms: Group B: Hip abductors strengthening exercises

SUMMARY:
The study will be a randomized controlled trial. Twenty-four subjects will be assigned randomly by using the lottery method into two groups. Group A will be given a hot pack in addition to the global hip muscles strengthening exercise while group B is the control group which will receive a hot pack in addition to hip abductor strengthening. The time duration will be 6 weeks. Pain intensity will be assessed by NPRS.3 sessions per week will be given for 6 weeks. Outcome measures will be taken at baseline, in 3rd week, and at the end of the 6th week.

DETAILED DESCRIPTION:
Secondary piriformis syndrome is a common condition of extra-spinal sciatica which is related to or around the piriformis muscle and irritates the sciatic nerve. Most cases reported are of secondary piriformis syndrome. Secondary piriformis syndrome is caused due to soft tissue inflammation, and muscular spasms, which result in nerve compression. Inflammation occurs due to trauma on the buttock and piriformis muscle contractures. Strengthening exercise program is another physical technique that has been supported by research in numerous areas, which has effects on the reduction of pain, range of motion, and lower extremity function. This study will aim to compare the effects of global hip muscles and isolated hip abductors muscle strengthening exercise programs on pain, range of motion, and lower extremity function in patients with secondary piriformis syndrome. The study will be a randomized controlled trial. Twenty-four subjects will be assigned randomly by using the lottery method into two groups. Group A will be given a hot pack in addition to the global hip muscles strengthening exercise while group B is the control group which will receive a hot pack in addition to hip abductor strengthening. The time duration will be 6 weeks. Pain intensity will be assessed by NPRS.3 sessions per week will be given for 6 weeks. Outcome measures will be taken at baseline, in 3rd week, and at the end of the 6th week. The collected data will be analyzed in the statistical package for the Social Sciences (SPSS) 25.Parametric/Non-parametric tests will be applied after testing the normality of the data.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* age: 20-50 years
* Batty test to diagnose secondary piriformis syndrome

Exclusion Criteria:

* Diagnosed Congenital spinal defects
* Diagnosed Hip arthritis
* Pregnancy
* Diagnosed Disc facet pathology
* History of Spinal trauma
* Musculoskeletal abnormality in the lumbar spine
* Diagnosed Rheumatologic disorders
* Any diagnosed bony or soft tissue systemic disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | follow up at 12th week
  Pain intensity will be assessed by NPRS. The 11-point NPRS (intervals from 0-10) isused to quantify pain intensity; 0 represents no pain, and 10 represent the worst possible agony. The NPRS is an valid and reliable instrument for older persons.Participants will be asked to select the number that most accurately describes theirlevel of pain. At the baseline assessment, following each exercise session during the12-week intervention, and finally at the end of the intervention Programme, the NPRS scores will be recorded.
Hand held dynamometer: | follow up at 12th week
  Using a Jamar hydraulic hand-held dynamometer, the isometric muscle strength ofthe involved hip abductor and extensor muscles will be measured (JHHD).
Goniometer: | follow up at 12th week
  The fulcrum and the body are placedover the joint being measured. The stationary arm is the arm of the goniometer thataligns with the inactive part of the joint measured. It is structurally a part of the bodyand is not movable independently of the body. The moving arm is the arm of the goniometer, which aligns with the mobile part of the joint measured.
Lower extremity function scale: | follow up at 12th week
  The LEFS can be used by clinicians as a measure of patients' initial function, ongoingprogress, and outcome as well as to set functional goals. LEFS to establish functionallevel, set goals, and track progress and outcome. Consider a patient with an initialLEFS score of 46/80. Based on the error at a given point in time for the LEFS of 5points, the clinician can be 90% confident that the actual scale score is between 41and 51. If the patient's condition is deemed to be relatively chronic and is expected tochange slowly, the clinician might select a 2-week time frame for a change in scoreof just at the MDC and MCID of 9 scale points. The short-term goal, therefore, couldbe: "Increase LEFS score to less than or equal to 54/ 80." In setting a short-term goalfor a patient with a relatively acute condition who is predicted to experience changequickly, a shorter time frame of, for example, 1 week with a greater change than theMDC and MCID may be selected

CONTACTS AND LOCATIONS:
Overall Officials: maria Abbas chishty, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah rehabilitation clinic, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwanaga J, Eid S, Simonds E, Schumacher M, Loukas M, Tubbs RS. The majority of piriformis muscles are innervated by the superior gluteal nerve. Clin Anat. 2019 Mar;32(2):282-286. doi: 10.1002/ca.23311. Epub 2018 Dec 21. PMID 30408241
- [Background] Cassidy L, Walters A, Bubb K, Shoja MM, Tubbs RS, Loukas M. Piriformis syndrome: implications of anatomical variations, diagnostic techniques, and treatment options. Surg Radiol Anat. 2012 Aug;34(6):479-86. doi: 10.1007/s00276-012-0940-0. Epub 2012 Feb 12. PMID 22327640
- [Background] Park JC, Shim JH, Chung SH. The effects of three types of piriform muscle stretching on muscle thickness and the medial rotation angle of the coxal articulation. J Phys Ther Sci. 2017 Oct;29(10):1811-1814. doi: 10.1589/jpts.29.1811. Epub 2017 Oct 21. PMID 29184293
- [Background] Filler AG. Piriformis and related entrapment syndromes: diagnosis & management. Neurosurg Clin N Am. 2008 Oct;19(4):609-22, vii. doi: 10.1016/j.nec.2008.07.029. PMID 19010285
- [Background] Shah SS, Consuegra JM, Subhawong TK, Urakov TM, Manzano GR. Epidemiology and etiology of secondary piriformis syndrome: A single-institution retrospective study. J Clin Neurosci. 2019 Jan;59:209-212. doi: 10.1016/j.jocn.2018.10.069. Epub 2018 Oct 24. PMID 30528358